CLINICAL TRIAL: NCT05720481
Title: Impact of Non Surgical Periodontal Treatment on Growth Differentiation Factor-15 Levels
Brief Title: Impact of Periodontal Treatment on Growth Differentiation Factor-15 Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Principal Investigator, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO-UniCt 125-2
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Root Planing

STUDY DESIGN:
Intervention Model Description: Each selected patient underwent randomly, without anaesthesia, after recording periodontal parameters, the two following treatments: in one, maxillary quadrants were treated as conventional Quadrant Scaling and Root Planing (SRP) or Full-Mouth Scaling and Root Planing
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis quadrant Scaling root planing (SRP) (Placebo Comparator): Each selected subject underwent to quadrant SRP
  Interventions: Other: Quadrant Scaling and root planing
- Periodontitis full mouth scaling root planing (SRP) (Active Comparator): Each selected subject underwent to full mouth SRP
  Interventions: Other: Full mouth Scaling and root planing

INTERVENTIONS:
Other: Full mouth Scaling and root planing — patients were treated with full mouth Scaling and root planing
  Arms: Periodontitis full mouth scaling root planing (SRP)
Other: Quadrant Scaling and root planing — patients were treated with quadrant Scaling and root planing
  Arms: Periodontitis quadrant Scaling root planing (SRP)

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence the management of Periodontitis, the aim of this study was to evaluates, at 6-months follow-up, the post-treatment clinical and serum parameters in patients with periodontitis, treated by either Full Mouth Scaling and Root Planing (FM-SRP) treatment versus conventional oral hygiene treatment on serum CRP and Growth differentiation factor-15 levels.

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2016. The local ethical committee approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent.

Subjects with a diagnosis of periodontitis were enrolled in this clinical trial. The inclusion criteria were: 1) good condition of general health, 2) a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm, 3) no involvement of the furcation, 4) a minimum of six teeth per quadrant, respectively. The exclusion criteria were: 1) periodontal therapy during the last 12 months, 2) assumption of antibiotics during the last 6 months, 3) pregnancy, 4) any systemic condition which might affect the effects of the study treatment, 5) previous or current radiation or immunosuppressive therapies, 5) use of mouthwash containing antimicrobials during the previous 3 months, 6) no use of hormonal contraceptives, 7) medication by anti-inflammatory and immunosuppressive drugs, 8) previous history of hard-drinking, 9) smoking, 10) class II and III tooth mobility. Patients randomly undergo to full mouth SRP or Quadrant SRP

ELIGIBILITY:
Inclusion Criteria:

* good condition of general health
* a minimum of 2 teeth for each quadrant with
* Pocket Depth (PD) ranging from 4-6 mm
* no involvement of the furcation
* a minimum of a six teeth per quadrant, respectively

Exclusion Criteria:

* periodontal therapy during the last 12 months
* assumption of antibiotics during the last 6 months
* pregnancy
* any systemic condition which might affect the effects of the study treatment
* previous or current radiation or immunosuppressive therapies
* use of mouthwash containing antimicrobials during the previous 3 months
* no use of hormonal contraceptives
* medication by anti-inflammatory and immunosuppressive drugs
* previous history of hard drinking
* smoking
* class II and III tooth mobility

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
reduction of Growth differentiation factor-15 serum levels | 6 months
  evaluation of serum Growth differentiation factor-15 change

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: Pubmed or internet

REFERENCES:
- [Derived] Isola G, Tartaglia GM, Santonocito S, Chaurasia A, Marya A, Lo Giudice A. Growth differentiation factor-15 and circulating biomarkers as predictors of periodontal treatment effects in patients with periodontitis: a randomized-controlled clinical trial. BMC Oral Health. 2023 Aug 21;23(1):582. doi: 10.1186/s12903-023-03237-y. PMID 37605193